CLINICAL TRIAL: NCT02011048
Title: Giant Ventral Incisional Hernia: Characteristics of Abdominal Muscle-matrix, and Effect of Hernia Repair on Abdominal Wall Function, Respiratory Performance and Quality of Life
Brief Title: Giant Ventral Incisional Hernia: Abdominal Wall Function, Respiratory Performance and Quality of Life
Acronym: GIVINA
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, PHD student, Bispebjerg Hospital
Other Study IDs: H-1-2013-097
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skeletal muscle biopsy, connective tissue biopsy, whole blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Giant ventral incisional hernia: Patient with a giant ventral incisional hernia (> 10 cm fascial defect) scheduled to undergo endoscopic components separation.
  Interventions: Procedure: Endoscopic components separation
- Control group: Patients scheduled to undergo surgery on other indications.

INTERVENTIONS:
Procedure: Endoscopic components separation — Endoscopic components separation hernia repair
  Groups: Giant ventral incisional hernia

SUMMARY:
One of five patients undergoing open abdominal surgery develops an abdominal wall defect (incisional hernia) as a late complication. A fraction of these are "giant" hernia with a fascial defect beyond 10 cm. These patients are physically severely impaired, and surgical treatment is complex.

Correction of giant incisional hernias including a relatively new and minimally invasive technique, (endoscopic components separation) offers promising results. This procedure allows the abdominal muscles to be joined centrally restoring the integrity of the abdominal wall.

The treatment of patients with giant hernia is now centralized at Bispebjerg Hospital allowing for a joint study between surgeons, pulmonologists, and sports medicine researchers to define the functional and biophysical outcome from hernia repair. We hypothesize that the abdominal muscle function is significantly optimized after restoration of the abdominal wall using this technique, and that muscular function is crucial for the postoperative quality of life. Moreover, we want to assess whether this operation specifically optimizes the function and protein synthesis of the abdominal wall muscles, and exerts a beneficial effect on lung function. Finally, we will investigate if the patients with giant incisional hernia may be identified by an altered composition of their connective tissue as compared with patients who do not develop incisional hernia.

This is a prospective study of two patient groups: 1) Patients with a giant incisional hernia and 2) controls undergoing open surgery on other indications. Assessment is done pre- and perioperatively and after 1 year including muscular function, lung function, abdominal wall anatomy as provided by CT-scan, and quality of life. Specified biopsies from muscles and connective tissue are examined for muscle fiber size/type and structure by various methods, including electron microscopy and atomic force microscopy. Lung function is monitored by blood gas concentrations, Chronic Obstructive Pulmonary Disease Assessment Test questionnaire, and regular spirometry analyses. The studies are carried out by Ph.D. student Kristian Kiim Jensen, and supervised by professor in surgery Lars Nannestad Jørgensen, professor in sports medicine Michael Kjær and professor in pulmonary medicine Vibeke Backer.

DETAILED DESCRIPTION:
Overall project aim

The present study examines the abdominal skeletal muscle and connective tissue of patients with giant ventral incisional hernia (VIH), and to evaluate the effect of a new endoscopic components separation technique (CST) with abdominal muscle replacement upon the muscular function of the abdominal wall and quality of life in patients. The study relies on the following hypotheses:

1. Collagen characteristics and organization are altered in patients with incisional hernia as compared with patients who do not develop incisional hernia.
2. Reconstruction of the linea alba by endoscopic CST and medialization of the abdominal rectus muscles in patients with giant VIH leads to improvement of daily function, respiratory performance and quality of life.
3. Abdominal wall reconstruction including CST with re-positioning of the rectus abdominis musculature increases the abdominal muscle mass and strength along with higher protein synthesis of the rectus muscles and a reduction of fibrotic skeletal muscle phenotype.

A total of 20 patients electively admitted for repair of a giant midline VIH, and 20 patients without hernias electively operated on for other indications are included. Exclusion criteria are pregnancy, severe heart- or lung disease, significant musculoskeletal disease, chemo- or radiotherapy within three months prior to the examination, and systemic corticosteroid medication. Oral and written informed consents are obtained from each participating patient.

Strength measurements of the m. rectus abdominis and the vastus lateralis of the quadriceps femoris muscle are done using a Good Strength muscle test system, both static and dynamic. The measurements are undertaken preoperatively and 1 year after surgery. A CT scan of the abdomen and thigh is done both 1 month before and 1 year after surgery to provide a detailed description of the hernia dimensions, the distance between the abdominal rectus muscles, and to determine the cross sectional area of the rectus abdominis and the vastus lateralis muscle. Lung function is determined by arterial blood gas, venous oxygen saturation, forced expiratory volume (FEV1), forced- and vital capacity (FVC, VC) including B2-receptor agonist reversal test, and maximum inspiratory- and expiratory pressure (MIP/MEP) preoperatively and 1 year postoperatively. Daily arterial blood gas is measured during postoperative admission. Lung function is determined at 1-month follow-up.

Quality of Life is assessed by the use of questionnaires. SF 36 is used for obtaining both mental and physical health scores. The St. George respiratory questionnaire and MRC are used to determine the level of daily lung impairment. Further, Carolina Comfort Scale assesses level of pain, movement limitation, and mesh sensation.

Protein turnover in both abdominal and thigh skeletal muscle is assessed by the use of a flood-primed continuous infusion of ring-13C6- phenylalanine. This will be infused four hours before surgery, and during this period 2-3 blood samples are drawn to verify stabilization of the isotope enrichment level prior to biopsy sampling. Muscle biopsy material is divided into fractions covering myofibrillar, sarcoplasmic and connective tissue proteins and analyzed using mass spectrometry to allow for calculation of protein synthesis of both contractile muscle protein and for muscle collagen. These procedures are repeated one year post surgery.

During surgery, biopsies of the linea alba, abdominal rectus muscle and the vastus lateralis muscle are taken using needle-biopsy equipment (Bergstrøm needle). One year after surgery the abdominal rectus muscle and vastus lateralis muscle again undergo the same biopsy procedure using a similar technique, but this time performed per-cutaneously under ultrasonographic guidance.

The biopsies are examined histologically for individual muscle fiber size and type (ATPase staining) as well as connective tissue and muscle structure (immunohistological examination collagen I, III and IV, laminin, desmin, tenascin-C). A section of the biopsy is used for mRNA expression by RT-PCR of COL1, COL3 and Tenascin-C. The content of collagen and both enzymatic and non-enzymatic cross-links (HP, LP and pentosidine) are determined by HPLC.

The linea alba connective tissue biopsy taken perioperative is investigated by electron microscopy for quantification of collagen fibril diameter, and atomic force microscopy to investigate fibril mechanics and 3-D structure of the connective tissue.

The change in abdominal flexor function and respiratory performance secondary to surgery is described in a paired design for both groups of patients. Quality of Life SF 36 and Carolina Comfort Scale are compared between the two groups of patients in an unpaired design and within patient groups in a paired design to assess any change induced by surgery. Differences between patient groups and change induced by surgery are assessed from the analyses on the harvested biopsy materials.

ELIGIBILITY:
Inclusion Criteria:

* Giant ventral incisional hernia with fascial defect > 10 cm
* Scheduled surgery on other indications
* Provided informed consent

Exclusion Criteria:

* Pregnancy,
* Severe heart- or lung disease
* Significant musculoskeletal disease
* Chemo- or radiotherapy within three months prior to the operation
* Systemic corticosteroid medication

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the outpatient clinic at Digestive Disease Center, Bispebjerg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Abdominal wall strength | Preoperative and one year postoperative
  Change in maximal abdominal wall strength measured by Good Strength system.

SECONDARY OUTCOMES:
Rectus abdominis muscle protein synthesis activity | Preoperative and one year postoperative
  The change in activity of the protein synthesis in rectus abdominis muscles of the patients.
Change in quality of life | Preoperative and one year postoperative
  Changes in quality of life measured by Carolinas Comfort Scale and SF-36
Change in respiratory function | Preoperatively, one month, and year postoperative
  Change in respiratory function as measured by spirometry and maximal inspiratory and expiratory pressure.
Maximal thigh strength | Preoperatively and one year postoperative
  Change in maximal thigh strength as measured by Power-Rig method.
Rectus abdominis muscle phenotype | Preoperatively and one year postoperative
  Changes in Rectus abdominis muscle phenotype due to hernia repair.
Connective tissue characteristics | Perioperatively
  Differences in connective tissue characteristics in patients with and without ventral incisional hernia.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nannestad Jorgensen, Dr. Msc, Study Chair — Digestive Disease Center, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen Northwest, Copenhagen, Denmark

REFERENCES:
- [Derived] Jensen KK, Oma E, Kjaer M, Jorgensen LN, Andersen JL. Histology and Function of the Rectus Abdominis Muscle in Patients With Incisional Hernia. J Surg Res. 2020 Sep;253:245-251. doi: 10.1016/j.jss.2020.03.033. Epub 2020 May 6. PMID 32387572
- [Derived] Jensen KK, Munim K, Kjaer M, Jorgensen LN. Abdominal Wall Reconstruction for Incisional Hernia Optimizes Truncal Function and Quality of Life: A Prospective Controlled Study. Ann Surg. 2017 Jun;265(6):1235-1240. doi: 10.1097/SLA.0000000000001827. PMID 27280505